CLINICAL TRIAL: NCT01279967
Title: A Randomized Stratified Multicentre Phase II Clinical Trial of Single Agent ADI-PEG 20TM (Pegylated Arginine Deiminase) in Patients With Malignant Pleural Mesothelioma
Brief Title: A Clinical Trial of ADI-PEG 20TM in Patients With Malignant Pleural Mesothelioma
Acronym: ADAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Cancer Research UK (Other); UK: Barts Center for Experimental Cancer Medicine (CECM) for Trial Coordination (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6837; 2006-004592-35 (EudraCT Number)
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2012-05

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Pleural Mesothelioma; ADI-PEG 20
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): Arm A is control arm with best supportive care.
- B (Experimental): Arm B is the treatment arm with best supportive care plus ADI-PEG20.
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20 — 36.8mg/m2 based on BSA, weekly treatment for 6 months
  Arms: B

SUMMARY:
To examine whether the arginine depleting drug, ADI-PEG 20, might be effective as a targeted therapy in patients with ASS-negative malignant pleural mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females aged 18 years and older. (There is no upper age limit)
2. Histopathological evidence of ASS-negative MPM. All biopsies will be reviewed for ASS expression using immunohistochemistry. Central lab confirmation is required before randomization
3. Performance status ECOG ≤ 1. Life expectancy should be greater than 3 months
4. Chemo-naive patients OR, Patients who have been previously treated with platinum-based combination chemotherapy with progressive disease at entry. In the event of a baseline diagnostic ASS-positive test, a repeat biopsy confirming loss of ASS expression will be required post platinum-based combination chemotherapy, with at least a 4 week interval from the last treatment episode.
5. CT evaluable disease by modified RECIST criteria
6. Adequate bone marrow function, or supported through treatment:

   * Haemoglobin 10g/dl or greater.
   * White cell count 2 x 109/L or greater, neutrophil count 1.5 x 109/L or greater
   * Platelets 75 x 109 /L or greater.
7. Adequate hepatic function (AST and ALT < 3 x upper limit of normal; bilirubin < 1.5 x upper limit of normal)
8. Creatinine clearance >30ml/min
9. Able to give written informed consent to participate

Exclusion Criteria:

1. Participation in another clinical trial using an investigational agent
2. Patients with surgically resectable disease
3. Recurrent pleural effusion (not pleurodesed)
4. Receipt of extensive radiation (hemi-thorax) therapy within 6 weeks before enrollment. Radiation to chest port sites following thoracotomy is permitted
5. A history of prior malignant tumour, unless the patient has been without evidence of disease for at least three years, or the tumour was a non-melanoma skin tumour or in-situ cervix carcinoma
6. Symptomatic or known brain or leptomeningeal metastases
7. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment
8. New York Heart Association (NYHA) Class III or IV heart failure (Attachment 10, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
9. Serious medical (e.g. uncontrolled diabetes, hepatic disease, infection, uncontrolled gout) or psychiatric illness likely to interfere with participation in this clinical study
10. History of seizures
11. Patients of child-bearing age must not become pregnant. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy. All patients enrolled on the study must agree to use acceptable birth control measures whilst on the study; using both barrier and hormonal methods. Patients that are surgically sterile are also eligible to participate in this study
12. Females must not be breastfeeding
13. Prior exposure to ADI-PEG 20
14. Preplanned surgery or procedures that would interfere with the study protocol
15. Allergy to pegylated products
16. Exposure to another investigational drug within 4 weeks prior to start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 18 months

SECONDARY OUTCOMES:
response rate | 18 months
overall survival | 18 months
time to progression | 18 months
safety (adverse events) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szlosarek, Principal Investigator — Barts and the London NHS
Locations (7):
- United Kingdom (7):
  - The Royal Sussex County Hospital, Brighton
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Hull and East Yorkshire Hospitals NHS Trust,The Princess Royal Hospital, Hull
  - Barts and The London NHS, St Bartholomew's Hospital, London
  - Guy's and St Thomas' Foundation Trust, Guy's Hospital, London
  - University Hospital of South Manchester NHS Foundation Trust, Wythenshawe Hospital, Manchester
  - Southampton University Hospitals NHS Trust, Southampton General Hospital, Southampton

REFERENCES:
- [Background] Szlosarek PW, Luong P, Phillips MM, Baccarini M, Stephen E, Szyszko T, Sheaff MT, Avril N. Metabolic response to pegylated arginine deiminase in mesothelioma with promoter methylation of argininosuccinate synthetase. J Clin Oncol. 2013 Mar 1;31(7):e111-3. doi: 10.1200/JCO.2012.42.1784. Epub 2013 Jan 14. No abstract available. PMID 23319692
- [Derived] Szlosarek PW, Steele JP, Nolan L, Gilligan D, Taylor P, Spicer J, Lind M, Mitra S, Shamash J, Phillips MM, Luong P, Payne S, Hillman P, Ellis S, Szyszko T, Dancey G, Butcher L, Beck S, Avril NE, Thomson J, Johnston A, Tomsa M, Lawrence C, Schmid P, Crook T, Wu BW, Bomalaski JS, Lemoine N, Sheaff MT, Rudd RM, Fennell D, Hackshaw A. Arginine Deprivation With Pegylated Arginine Deiminase in Patients With Argininosuccinate Synthetase 1-Deficient Malignant Pleural Mesothelioma: A Randomized Clinical Trial. JAMA Oncol. 2017 Jan 1;3(1):58-66. doi: 10.1001/jamaoncol.2016.3049. PMID 27584578
- See also: Related Info — http://www.cancer.qmul.ac.uk/staff/szlosarek.html